CLINICAL TRIAL: NCT01053832
Title: Ventricular Pace Suppression Study With the EVIA/ENTOVIS DR-T/DR Pacemaker
Brief Title: Ventricular Pace Suppression Study
Acronym: VpS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 45
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Pacemaker Indication
Keywords: ventricular pace suppression; pacemaker; efficacy; safety; support of intrinsic heart rhythm

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Ventricular Pace Suppression- ON (Other)
  Interventions: Device: VpS algorithm in EVIA and ENTOVIS pacemakers
- Ventricular Pace Suppression- OFF (Other)
  Interventions: Device: VpS algorithm in EVIA and ENTOVIS pacemakers

INTERVENTIONS:
Device: VpS algorithm in EVIA and ENTOVIS pacemakers — For one group of patients, the VpS algorithm will be activated and for the other group, the VpS algorithm will be deactivated until the cross-over, where these conditions will be switched.

SUMMARY:
Investigation of the efficacy and safety of the Ventricular Pace Suppression (VpS) algorithm.

DETAILED DESCRIPTION:
The aim of this study is to investigate the percentage of reduction of ventricular pacing using the VpS feature of the EVIA/ENTOVIS pacemaker in a controlled clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal AV block and/or Sinus Node Dysfunction
* DDD(R)-ADI(R)-Mode (VpS Algorithm) applicability

Exclusion Criteria:

* Permanent AV block III°
* Permanent Atrial Fibrillation/ Flutter
* Require mode other than DDD(R)-ADI(R) or DDD(R)
* Have a life expectancy of less than six months
* Expected to receive heart surgery within six months
* Enrolled in another cardiac investigation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Reduction of right ventricular pacing with the help of the VpS algorithm in the EVIA/ ENTOVIS pacemakers. | 6-8 months

SECONDARY OUTCOMES:
A Complication free rate >95%, with respect to the VpS feature of the implanted pacemaker. | 6-8 months

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Bonnemeier, Prof. Dr., Principal Investigator — Klinik für Kardiologie und Angiologie, UNIVERSITÄTSKLINIKUM Schleswig-Holstein, Campus Kiel
Locations (2):
- Germany (2):
  - Klinikum Coburg gGmbH, Coburg, Bavaria
  - Abteilung für Elektrophysiologie, Klinik für Kardiologie und Angiologie, UNIVERSITÄTSKLINIKUM Schleswig-Holstein, Kiel, Schleswig-Holstein